CLINICAL TRIAL: NCT02838771
Title: Validation and Clinical Application of Dysphagia Screening Questionnaire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Collaborators: Klaipėda University (Other)
Responsible Party: Principal Investigator, Nora Siupsinskiene, Professor medical doctor of otorhinolaryngology, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DSQ1
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2013-12

CONDITIONS: Dysphagia; Swallowing Disorders
Keywords: Swallowing Disorder; Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Research group participants (Experimental): Research group consisted of 171 elderly nursing home residents and 82 outpatients of the Hospital of Lithuanian University of Health Sciences.
  The participants were given the dysphagia screening questionnaire, consisted of 16 questions and the several sips of water to drink (clinical water drinking test for dysphagia screening).
  Interventions: Other: Water drinking test; Other: Dysphagia screening questionnaire
- Control group participants (Other): Community-dwelling elderly healthy individuals. The participants were given the dysphagia screening questionnaire, consisted of 16 questions and the several sips of water to drink (clinical water drinking test for dysphagia screening).
  Interventions: Other: Water drinking test; Other: Dysphagia screening questionnaire

INTERVENTIONS:
Other: Water drinking test — Patient takes a sip of water about 60-70 ml. We assess: coughing, choking, voice changes.
Other: Dysphagia screening questionnaire — Lithuanian version of the questionnaire consists of 16 questions. Interpretation of dysphagia screening questionnaire: advanced symptom - 2 points, moderate intensity symptom - 1 point, no symptom - 0 point. At least one advanced symptom means - dysphagia. Higher score represents stronger dysphagia intensity. The maximum score is 32 points.

SUMMARY:
The aim of this research was to develop a dysphagia screening measure and evaluate the prevalence of dysphagia and its clinical manifestation in different in age population groups.

DETAILED DESCRIPTION:
The dysphagia screening questionnaire had the stages of validation - translation and back translation, a review of the translation and back translation committee, pre-test study (36 persons) with monolingual individuals and the test re-test study (67 subjects included).

The case - control study groups were tested using dysphagia screening questionnaire and clinical screening - water drinking test. Barthel index and nutrition questionnaire were used to identify the nutritional and functional state. M. D. Anderson dysphagia inventory questionnaire, sf-12 questionnaire were used to assess dysphagia effects on the quality of life.

The research group consisted of two subgroups - 171 nursing home residents from 3 different nursing homes and 82 outpatients of the Hospital of Lithuanian University of Health Sciences. The control group consisted of randomly selected 40 community-dwelling elderly healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Consent for participating in the research
* No cognitive disorders or mental illnesses

Exclusion Criteria:

* Refusal to participate in the research
* Serious mental or cognitive conditions

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 293 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Dysphagia screening questionnaire | At the baseline
  Lithuanian version of questionnaire consists of 16 questions about masticatory and swallowing functions and dysphagia consequences during patients last one year.

SECONDARY OUTCOMES:
Clinical water drinking test | At the baseline
  A subject takes one tablespoon of water. Then - a sip of water (about 60-70 ml). We assess: coughing, choking, voice changes. At least one symptom means dysphagia.
Barthel index | At the baseline
  Barthel index was used to identify objectively the functional state. According to Barthel index 100 points mean - functional independency, 91 - 99 - little dependency, 61 - 90 - moderate dependency, 21 - 60 - almost total dependency, 0 - 20 - total dependency.
Nutrition questionnaire | At the baseline
  Nutrition questionnaire was used to identify objectively the nutritional state. The maximal score of nutritional state questionnaire - 30. 24 or more points mean - good nutritional state, 17-23,5 - risk of insufficient nutrition, < 17 - insufficient nutrition.
M. D. Anderson dysphagia inventory (MDADI) | At the baseline
  Assessment if dysphagia effects the quality of life. Questionnaire consists of 20 questions. The emotional, functional, physical and global subscales are measured. Scores of each item can be from 0 to 100, they are summed, a mean score is calculated. A higher MDADI score represents better functioning and better quality of life.
The 12-Item Short Form Health Survey (SF-12 questionnaire) | At the baseline
  Assessment of the quality of life, general health status using 12 questions. Assess physical functioning, role limitation due to physical problems, bodily pain, general health, vitality, social functioning, limitations in usual role activities because of emotional problems, mental health. Scores range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Siupsinskiene, Professor, Principal Investigator — Lithuanian University of Health Sciences Otorhinolaryngology department; Nora Siupsinskiene, Professor, Principal Investigator — Klaipėda University
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided